CLINICAL TRIAL: NCT06385743
Title: The Effectiveness of Neuromuscular Training-Based Exercise Program Among Overhead Athletes With Shoulder Pain
Brief Title: The Effectiveness of Neuromuscular Training-Based Exercise Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Principal Investigator, Asli Yeral, Physiotherapist, MSc. (principal Investigator), Yeditepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: yeditepe15
Record Dates: First submitted 2023-04-10; First posted 2024-04-26 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Pain, Shoulder; Sports Physical Therapy
Keywords: Overhead Athletes; Neuromuscular training; Shoulder funtions; Shoulder pain; performance
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular Training-based Exercise Program Group (Experimental): Patient Education: Both groups will be given patient education on pain mechanism, posture/posture, exercise training, the role of the shoulder joint in shooting mechanics, situations, and positions to be avoided.
  Neuromuscular Training-based Exercise Program: This group will be given a neuromuscular training-based exercise program in a total of 24 physiotherapy sessions, 3 days a week, for eight weeks. In addition to shoulder strength, stabilization and kinetic chain exercises, this program includes internal and external focus (sound, touch, light, dual task, etc.), sport-specific exercises and plyometric exercises (speed, agility).
  Interventions: Other: Neuromuscular Training-based Exercise Program
- Thrower's Ten Exercise Program Group (Active Comparator): Patient Education: Both groups will be given patient education on pain mechanism, posture/posture, exercise training, the role of the shoulder joint in shooting mechanics, situations, and positions to be avoided.
  Thrower's Ten Exercise Program: This group will be given include Thrower's Ten Exercise Program in a total of 24 physiotherapy sessions, 3 days a week, for eight weeks. This program includes 10 different shoulder strengthening and shoulder stabilization exercises in a diagonal pattern. "Advanced Thrower's Ten" exercises that include kinetic chain exercises (covering more than one joint) in addition to shoulder exercises planned to be used in the late stages of rehabilitation into the program, progression is considered after the 3rd week will be added.
  Interventions: Other: ''Thrower's Ten'' Exercise Program

INTERVENTIONS:
Other: Neuromuscular Training-based Exercise Program — Neuromuscular training has been accepted as an effective treatment modality to improve the neurophysiological states of the joints for coordinated work. In addition to shoulder strength, stabilization and kinetic chain exercises, this program includes internal and external focus (sound, touch, light, dual task, etc.), sport-specific exercises and plyometric exercises (speed, agility). All athletes with shoulder pain will include in the baseline evaluation at the beginning of the season and all parameters will be followed throughout the season for 8 weeks. All athletes in this group will participate in a total of 24 physiotherapy sessions, 3 days a week, for eight weeks.
  Arms: Neuromuscular Training-based Exercise Program Group
Other: ''Thrower's Ten'' Exercise Program — ''Thrower's Ten'' Exercise Program includes 10 different shoulder strengthening and shoulder stabilization exercises in a diagonal pattern. "Advanced Thrower's Ten" exercises that include kinetic chain exercises (covering more than one joint) in addition to shoulder exercises planned to be used in the late stages of rehabilitation into the program, progression is considered after the 3rd week will be added. All athletes with shoulder pain will include in the baseline evaluation at the beginning of the season and all parameters will be followed throughout the season for 8 weeks. All athletes in this group will participate in a total of 24 physiotherapy sessions, 3 days a week, for eight weeks.
  Arms: Thrower's Ten Exercise Program Group

SUMMARY:
This randomised controlled study aimed to investigate the effectiveness of a neuromuscular training-based exercise program on pain, function, risk factors specific to shoulder injuries and performance in overhead athletes with shoulder pain.

The main hypothesis is;

H0: There is no difference between the "Thrower's Ten" exercise program and the neuromuscular training-based exercise program applied to overhead athletes with shoulder pain, on pain, function, risk factors specific to shoulder injuries, and performance.

H1: The effects of a neuromuscular training-based exercise program on pain, function, risk factors specific to shoulder injuries and performance in overhead athletes with shoulder pain are superior to the effects of "Thrower's Ten" exercise program

DETAILED DESCRIPTION:
Overhead athletes with shoulder pain who met the inclusion criteria applied to Yeditepe University Hospital Orthopedics and Traumatology Clinic for a randomized controlled study will be included to demonstrate the effectiveness of a neuromuscular training-based exercise program in overhead athletes with shoulder pain.

Athletes will be included in two different exercise programs (Thrower's Ten and Neuromuscular Training Based groups) by simple randomization.

Athletes evaluated by the orthopaedic surgeon will be included in the study if willing to participate in the rehabilitation program. The treatment program to be applied, hands-off treatment, was determined as exercise therapy. In our study, the athletes participating in the Neuromuscular Training-Based Exercise Program (Group 1) and the ''Thrower's Ten'' Exercise Program (Group 2) will participate in 24 physiotherapy sessions, three days a week, for eight weeks.

Before starting the treatment program, the participants' sociodemographic characteristics, comorbidities, dominant sides, sports histories, training routine (frequency/week, duration, etc.), and previous injury histories will be questioned with a structured evaluation form. Before randomization, a clinical examination for shoulder pain will be done by the orthopaedic surgeon. Pain intensity, pressure pain threshold, muscle tone, shoulder functional status, risk factors specific to shoulder injuries, sportive performance and kinesiophobia will be evaluated before treatment, at the end of the eight-week exercise program,

ELIGIBILITY:
Inclusion Criteria:

* Giving consent to be a volunteer for participating
* 18-35 years of age
* Athletes playing overhead sports like volleyball, water polo, tennis, baseball, cricket, swimming, badminton, and basketball for at least 2 days a week (Unilateral sports).
* Patients with unilateral shoulder pain lasting >6 weeks.
* Suitable and referred for conservative treatment by an orthopedist (non-surgical patients)
* Having one positive sign in the following 3 categories; the painful arc of movement, Neer or Hawkins-Kennedy impingement signs and pain during resisted external rotation, abduction, or empty can test performed by the orthopedist.
* Participating in regular training with the team for at least 3 years of experience in overhead sports

Exclusion Criteria:

* Bilateral shoulder pain
* Having an acute shoulder pain
* Having a non-specific shoulder pain
* Reflected pain
* Having some severe shoulder patholojies such as adhesive capsulitis, osteoarthritis, rheumatoid arthritis, fracture, dislocation and instability
* Shoulder pain originating from non-musculoskeletal system
* Having the shoulder and neck surgery and non-traumatic injuries within the last six months
* Having severe pathologies during the rehabilitation program (cardiac, diabetes mellitus and neuropsychiatric problems)
* Presence of diagnosed significant comorbidity (neurological and systemic disorders)
* Current and past carcinoma
* Type 3 acromion
* Avulsion fracture
* Non-compliance with treatment
* Symptomatic cervical spine pathology
* Antidepressant usage
* Clinical signs of full-thickness rotator cuff tears (positive lag signs)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Pain Assessment | 8 weeks
  Visual Analogue Scale will be used to evaluate the severity of pain felt around the shoulder joint. The location of the pain and the severity of the pain will be questioned. Participants will be asked to indicate pain severiy they felt (rest, activity and night) on a 10 cm horizontal line, ranging from 0 to 10. Zero shows no pain and 0 is intolerable pain. Pain intensity will be recorded by measuring the value of the marked place in cm. Higher values indicate more severe pain.
Disabilities of the Arm, Shoulder and Hand (DASH) | 8 weeks
  The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire was used to evaluate status of shoulder function. It is a questionnaire that evaluates all upper extremity functions and consists of a total of thirty questions. 21 of the questions of the questionnaire question the ability to perform functional activities, 5 of them about pain and 4 of them about the psychosocial effects of the disease. Each question is scored using a 5-point Likert scale with a range of 1-5. The total score of the questionnaire varies between 0-100 points, higher scores indicate better functional status. DASH, which has a short completion time and moderate scoring ease, is a questionnaire that can be used in patients between the ages of 18-64.

SECONDARY OUTCOMES:
Tampa Kinesiophobia Scale | 8 weeks
  Tampa Kinesiophobia Scale (Tampa Kinesiophobia Scale, TKS) was used for kinesiophobia. TKS is a 17-item scale consisting of questions about re-injury anxiety, pain, anxiety, and fear-avoidance behaviors. This questionnaire is used for diseases associated with chronic and acute pain, musculoskeletal injuries and fibromyalgia. This scale utilizies a 4-point Likert score with 1-4 intervals (1= Strongly disagree, 4 = Strongly agree).
Hylyght Injury Prevention and Return to the Sports Screening Program ( | 8 weeks
  This program will be used to evaluate risk factors specific to shoulder pain in overhead athletes. The physiotherapist will evaluate each athlete using these specific shoulder injury risk factors tests, and the results will be recorded in the system. These risk factors include parameters for the shoulder (flexibility, strength, range of motion, core stability). The application will automatically generate an individual risk profile map showing risk levels in red, yellow, and green based on AI according to the category of the entered value. Database will be determined pain specific risk factors according to prospective studies. Each participant's individual risk profile will be formed.Both groups' risk profile map changes before and after treatment will be evaluated.
Y Balance Test- Upper Quarter | 8 weeks
  Upper Quarter Y-Balance Test (UQYBT) which is a functional performance test will be used to evaluate kinetic chain, mobility, and stability the components of upper extremity in a closed kinetic chain. The YBT-UQ which is called a closed kinetic chain functional screening tool with using the Y Balance Test kit (Move2Perform, Evansville, IN, USA). Participants will be positioned push-up position with the center of one hand on the grid. Participants will reach out as far as possible in the tested direction. Physiotherapist will measure the reach distance expressed in refrence to the stance limb which is tested side.
Closed Kinetic Chain Extremity Stability Test | 8 weeks
  Closed Kinetic Chain Extremity Stability (CKCUES) Test was applied to participants with shoulder dysfunctions and to assess shoulder performance. Athletes will be positioned in push- ups position between tapes. Athletes will move their hands back and forth, touching each tape. The physiotherapist will count the athlete's touch number within 15 seconds.
Single Arm Seated Shot Put Test | 8 weeks
  The Single Arm Seated Shot Put Test (SSPT) is defined as an upper extremity functional performance test used in the clinical setting. In the test, a weighted ball is asked to be pushed forward during a shooting motion. Few pieces of equipment are requaried for this test. Physiotherapists will be positioned athletes to sit upright with the back, pelvis, shoulders, and head against the wall. Other hand will be resting on the floor or on the lap. Athletes will shot- put the ball as far as possible without moving away from the wall. The physiotherapist will measure where the ball first struck the ground for all three attempts in centime.

CONTACTS AND LOCATIONS:
Overall Officials: Aslı Yeral, MSc, Principal Investigator — Yeditepe University
Locations (1):
- Yeditepe University, Istanbul, Turkey (Türkiye)